CLINICAL TRIAL: NCT02556281
Title: PROGNOSTIC VALUE OF CIRCULATING TUMORAL FREE DNA Versus CIRCULATING TUMORAL CELLS IN PATIENTS WITH COLORECTAL CANCER STAGE II-III
Acronym: CTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/066/HP
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with colorectal cancer (Experimental): Blood sampling is done for patient with colorectal cancer
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood sampling is done for patient with colorectal cancer

SUMMARY:
After curative surgical resection, detection of metastatic lymph node remains the main prognostic validated criteria on which is based the decision of adjuvant therapy. To date, none of the molecular alterations, identified as potentially predictive factor, are used in routine for therapeutic decision. The circulating markers, either in the form of free circulating DNA or in the form of circulating tumoral cells seems important potential candidates. To investigators knowledge, only one study estimated with several interesting results the prognostic interest of a coupled detection of the free circulating mutant DNA (gene KRAS) and by the hypermethylation of the p16 gene. Definitive conclusions remain however difficult to achieve because of the small number of patient included (n=58) and the fact that this study included different stages. For colorectal cancer a Chinese team presented a series of results suggesting that the presence of CTC during the postoperative course is a factor significantly related to the risk of recurrence. In multivariate analysis integrating the lymph node status and the vascular invasion, the presence of CTC appeared as an independent factor for recurrence with a hazard ratio of 29.5.

The aim of the present study is to compare the prognostic value of two circulating tumoral markers KRAS point mutations and RASSF2A methylation (free tumoral DNA) and Circulating tumoral cells (CTC). The primary objective is to compare sensibility and specificity of two circulating markers (free tumoral DNA and tumoral cells) on 2 years disease free survival rate. Secondary objective is to confirm the prognostic value of circulating free tumoral DNA and circulating tumoral cells in localised colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age superior to 18 years.
* Histologically confirmed colonic or rectal adenocarcinoma.
* stage II or III (TNM classification).
* Curative resection (R0)
* Absence of metastasis (abdominal ultrasonography or CTscan and pulmonary Rx or CTscan) in exams performed within 4 weeks.
* ECOG performance status <3.
* Signed and dated informed consent document.

Exclusion Criteria:

* Metastatic disease.
* Familial adenomatous polyposis
* Prior chemotherapy and or radiotherapy within 6 weeks
* Medical history of cancer within 5 years except: basocellular cutaneous neoplasia and intraepithelial neoplasia of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2012-10-15 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Presence of free tumoral DNA in blood of patient with colorectal cancer | Day 1
  Presence of free tumoral DNA (yes/no) in blood of patient with colorectal cancer
Number of patient with a first relapse | 24 Months
  Number of patient with a first relapse, defined by discovering of new lesion or metastasis

SECONDARY OUTCOMES:
Presence of tumoral cells in blood of patient with colorectal cancer | Day 1
  Presence of tumoral cells (yes/no) in blood of patient with colorectal cancer
Number of tumoral cells in blood of patient with colorectal cancer | Day 1
  Quantification of tumoral cells in blood of patient with colorectal cancer
Number of free tumoral DNA in blood of patient with colorectal cancer | Day 1
  Quantification of free tumoral DNA in blood of patient with colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jean J TUECH, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France